CLINICAL TRIAL: NCT06397677
Title: Defining the Molecular and Radiologic Phenotype of Progressive RA Interstitial Lung Disease (MOUNTAIN)
Brief Title: Defining the Molecular and Radiologic Phenotype of Progressive RA Interstitial Lung Disease
Acronym: MOUNTAIN
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of California, San Francisco (Other); University of Michigan (Other); University of Kansas (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0295; 1R01HL168126-01 (NIH)
Record Dates: First submitted 2023-12-01; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial | interventions — Laboratories

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Blood will be obtained for DNA (deoxyribonucleic acid), RNA (ribonucleic acid), serum, and plasma at baseline and at 12 months for all sites. For subjects enrolled in the study at the University of Colorado, peripheral blood samples will be obtained every 3-4 months. Samples not being directly assayed will be banked for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with RA-ILD: Assessments include:
  * Clinical: height, weight, oxygen saturation at rest, and 6-minute walk test.
  * Rheumatological: study Rheumatologist will document rheumatoid arthritis symptoms and clinical findings at baseline and follow-up.
  * Pulmonary Function Testing: data will be collected from clinically performed spirometry and diffusing capacity for carbon monoxide.
  * High-resolution computed tomography (HRCT) imaging: HRCT scans will be collected at baseline and 12 months in line with standard of care for treatment of RA-ILD.
  * Lab specimens: peripheral blood will be obtained for DNA, RNA, serum, and plasma at baseline and at 12 months for all sites or every 3-4 months in Colorado. Buccal swabs (cheek) will also be collected once each year.
  * Information collected: will include demographics, co-morbidities, disease history, medication history, pulmonary function, radiographic imaging, and transplant/survival status through questionnaires and medical chart review.
  Interventions: Genetic: Research Testing Performed (Laboratory); Diagnostic Test: Information Collected as Standard of Care; Other: Research Testing Performed

INTERVENTIONS:
Genetic: Research Testing Performed (Laboratory) — Blood collection (DNA, RNA)
Diagnostic Test: Information Collected as Standard of Care — High Resolution CT Scan (Chest), Pulmonary Function Testing (PFT), 6-Minute Walk Test (6MWT)
Other: Research Testing Performed — Blood collection (non-genetic), Buccal Swab, Rheumatologic Assessment, Pulmonary Assessment, Questionnaires

SUMMARY:
A study to identify patients with Rheumatoid Arthritis - Associated Interstitial Lung Disease (RA-ILD) that are at the highest risk for progression.

The goal of the investigators is to recruit a group of patients with RA-ILD and collect information to help us understand more about disease progression. The investigators will do this using a combination of clinical, radiologic, and biologic features.

DETAILED DESCRIPTION:
The central hypothesis is that novel quantitative imaging and specific blood markers will be associated with progressive RA-ILD. The hypothesis will be tested through collection and analysis of peripheral blood, in addition to the analysis of HRCT (high-resolution computed tomography) scans performed as standard of care (clinical) on research subjects.

Procedures performed:

Baseline Year 0: Blood sample, buccal (cheek) swab, questionnaires and if performed clinically - Pulmonary Function tests, 6 Minute Walk Test, and HRCT scan of lungs

Every 4 months (at clinic visit): Blood sample, questionnaires

Year 1 and Year 2 Follow-ups: Blood sample, buccal (cheek) swab, questionnaires and if performed clinically - Pulmonary Function tests, 6 Minute Walk Test, and HRCT scan of lungs

ELIGIBILITY:
Inclusion Criteria:

* Multidisciplinary diagnosis of RA-ILD based on the 2010 American College of Rheumatology criteria
* 18 years of age or older

Exclusion Criteria:

* Prior medication treatment specifically for RA-ILD
* Inability to give informed consent
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA-ILD study patients will be recruited from the University of Colorado Hospital, ILD Clinic (CU, PI: Joyce Lee, MD), in addition to the Rheumatology Clinic at the University of Colorado Hospital. Subjects will additionally be recruited from three unaffiliated ILD centers: University of California San Francisco (UCSF; site PI Dr. Paul Wolters), University of Kansas (KU, site PI Dr. Scott Matson), and University of Michigan (UM, site PI Dr. Justin Oldham).
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating the role of novel quantitative imaging | 5-years
  Through evaluation of baseline CT scans and application of novel quantitative technology, investigators will monitor for specific patterning to identify patients at risk for progression.

SECONDARY OUTCOMES:
Comparing peripheral blood telomere length (PB-TL) | 5-years
  Investigators will test and validate if baseline peripheral blood telomere length (PB-TL) predicts a progressive phenotype in RA-ILD.
Defining peripheral blood transcriptomic profiles | 5-years
  Investigators will define and validate the peripheral blood transcriptomic profile of progressive RA-ILD.
Exploring if a composite profile more accurately identifies progressive RA-ILD | 5-years
  Investigators will use logistic least absolute shrinkage and selection operator (LASSO) to develop a predictive model of RA-ILD progression using demographics, novel imaging, PB-TL and peripheral blood transcriptome.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce S Lee, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Kansas, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No